CLINICAL TRIAL: NCT03379779
Title: Department of Critical Care Medicine, Taichung Veterans General Hospital
Brief Title: Evaluation the Association of Microbiome Between Respiratory Tract Samples and Stool Samples in Pneumonic Patients Accompanied by Respiratory Failure
Status: Completed | Type: Observational
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Principal Investigator, Pin-Kuei Fu, MD, PhD, Principal Investigator, Department of Critical Care Medicine, Taichung Veterans General Hospital
Other Study IDs: IGA-10601
Record Dates: First submitted 2017-12-14; First posted 2017-12-20 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Microbiota; Pneumonia, Bacterial; Respiratory Failure; Lower Resp Tract Infection
Keywords: Microbiota; Respiratory Failure; Pneumonia; Lower Respiratory Tract Infection
MeSH Terms: conditions — Pneumonia, Bacterial; Respiratory Insufficiency; Pneumonia | interventions — Defecation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Blood sample obtained for cytokines detection
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pneumonia patient with respiratory failure: Sputum and stool sampling day 1, 3 and 7 after enrolling into study
  Interventions: Diagnostic Test: 16s RNA sequence of sputum, bronchoalveolar lavage fluid (options), stool

INTERVENTIONS:
Diagnostic Test: 16s RNA sequence of sputum, bronchoalveolar lavage fluid (options), stool — We will check the microbiome in lower respiratory samples (sputum and bronchoalveolar lavage fluid) and stool by using 16S RNA sequencing

SUMMARY:
A prospective observational study. Enrolled participants admitted to ICU due to pneumonia and respiratory failure need mechanical ventilator support. Investigators collected the residual specimens, such as sputum from endotrachea aspiration, bronchoalveolar lavage fluid in those participants as the usual care in the ICU. Those residual samples were sent to extract RNA and sequence by using high-throughput sequencing (next-generation sequencing) method.

Investigators will compared the microbiome feature between lower respiratory tract and stool specimens in those participants diagnosed as pneumonia with respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged than 40 years old
* Diagnosed as pneumonia
* Respiratory failure with mechanical ventilator support

Exclusion Criteria:

* Less than 40 years old
* Has been treated with antibiotics more than 7 days within two weeks before enrolling into study
* Suspected or active pulmonary tuberculosis infection

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who suffered from pneumonia and respiratory failure needed mechanical ventilator support with inform consent will be enrolled into study
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
The dynamics of the airway bacterial microbiome in the lower respiratory tract specimens in the setting of pneumonia accompanied by respiratory failure at the onset of, and day 3 and day 7 (or before extubation) | Compared the dynamic change of mirobiome at the baseline (onset of respiratory failure within 48 hours)m day 3 and day 7
  Uses high-throughput sequencing (next-generation sequencing) to sequence the 16S rRNA sequence of bacteria in residual samples

SECONDARY OUTCOMES:
The dynamics of the gut bacterial microbiome in the stool specimens in the setting of pneumonia accompanied by respiratory failure at the onset of, and day 3 and day 7 (or before extubation) | Compared the dynamic change of mirobiome at the baseline (onset of respiratory failure within 48 hours)m day 3 and day 7
  uses high-throughput sequencing (next-generation sequencing) to sequence the 16S
The association of the microbiome between lower respiratory tracts and stool specimens in pneumonic patient with respiratory failure | Compared the association of mirobiome at the baseline (onset of respiratory failure within 48 hours)m day 3 and day 7
  Uses high-throughput sequencing (next-generation sequencing) to sequence the 16S

CONTACTS AND LOCATIONS:
Overall Officials: Pin-Kuei Fu, MD, PhD, Principal Investigator — Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
We will share study protocol and Informed Consent Form and Clinical Study Report to other researchers
Supporting Information: Study Protocol, ICF, CSR
Time Frame: One year after the study was completed
Access Criteria: E-mail to yetquen@gmail.com Dr. Pin-Kuei Fu